CLINICAL TRIAL: NCT04385875
Title: Study to Assess the Safety and Durability of Viral Control Beyond 24 Weeks of Analytical Treatment Interruption After the Administration of Candidate HIV-1 Vaccines DNA.HTI, MVA.HTI and ChAdOx1.HTI or Placebo in Early Treated HIV-1 Positive Individuals (ATI Extension of AELIX-002 Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Aelix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ATI_extension
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infection; Therapeutic Vaccines; HTI; Antiretroviral Treatment Interruption (ATI); Viral control
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: Participants of the AELIX-002 clinical trial were randomly allocated to one of the following arms:
  * Vaccine: DNA.HTI at weeks 0, 4, and 8 and MVA.HTI at weeks 12 and 20 (DDDMM) followed by ChAdOx1.HTI at weeks 0 and 12 and MVA.HTI at week 24 (CCM), starting at least 24 weeks after MVA.HTI week 20.
  * Placebo: Normal saline solution at weeks 0, 4, 8, 12, and 20 (PPPPP) followed by normal saline solution at weeks 0, 12 and 24 (PPP), starting at least 24 weeks after week 20 administration.
  ATI_extension will keep allocation from AELIX-002 for a separate description of the results.
Who Masked: Participant, Investigator
Masking Description: AELIX-002 was a double-blind clinical trial. During ATI_extension, AELIX-002 will be unblinded and allocation will be disclosed to both participants and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine group (Experimental): ATI_extension will keep allocation from AELIX-002 for a separate description of the results.
  Interventions: Biological: Vaccine + extension of the ATI period
- Placebo group (Placebo Comparator): ATI_extension will keep allocation from AELIX-002 for a separate description of the results.
  Interventions: Other: Placebo + extension of the ATI period

INTERVENTIONS:
Biological: Vaccine + extension of the ATI period — During the AELIX-002 trial participants received the following: DNA.HTI at weeks 0, 4, and 8 and MVA.HTI at weeks 12 and 20 (DDDMM) followed by ChAdOx1.HTI at weeks 0 and 12 and MVA.HTI at week 24 (CCM), starting at least 24 weeks after MVA.HTI week 20. After that, on ATI_extension trial, ATI will be extended for 48 weeks.
  Arms: Vaccine group
Other: Placebo + extension of the ATI period — During the AELIX-002 trial participants received the following: Normal saline solution at weeks 0, 4, 8, 12, and 20 (PPPPP) followed by normal saline solution at weeks 0, 12 and 24 (PPP), starting at least 24 weeks after week 20 administration. After that, on ATI_extension trial, ATI will be extended for 48 weeks.
  Arms: Placebo group

SUMMARY:
The AELIX-002 trial has been conducted on a cohort of individuals who started cART within the first 6 months after the primary VIH infection, thus increasing the likelihood of observing a certain rate of post-treatment controls (PTC), regardless of treatment efficacy. Although the kinetics of HIV rebound should allow observing differences between placebo and control regarding the post treatment controls rate in case of efficacy of the IMPs, assessing the length and determinants of a post-intervention control (PIC) (i.e., associated with vaccination) beyond 24 weeks is crucial for developing a curative approach to HIV infection. In this regard, an extension of the ATI phase for those individuals with pVL less than 2,000 copies/mL after 24 weeks of ATI in the AELIX-002 offers an unique research opportunity to better understand relevant aspects of the mechanisms involved in the different phenotypes of a PIC and PTC.

DETAILED DESCRIPTION:
The AELIX-002 trial has been conducted on a cohort of individuals who started cART within the first 6 months after the primary VIH infection, thus increasing the likelihood of observing a certain rate of post-treatment controls (PTC), regardless of treatment efficacy. Although the kinetics of HIV rebound should allow observing differences between placebo and control regarding the post treatment controls rate in case of efficacy of the IMPs, assessing the length and determinants of a post-intervention control (PIC) (i.e., associated with vaccination) beyond 24 weeks is crucial for developing a curative approach to HIV infection. In this regard, an extension of the ATI phase for those individuals with pVL less than 2,000 copies/mL after 24 weeks of ATI in the AELIX-002 offers an unique research opportunity to better understand relevant aspects of the mechanisms involved in the different phenotypes of a PIC and PTC.

This trial will enrol participants of the AELIX-002 clinical trial regardless of whether they received vaccines or placebo, who reach 24 weeks of ATI with pVL <2,000 cop/ml and are willing to remain off cART. After accepting participation, subjects will undergo a one-year extension [48 weeks] of ATI monitoring (total duration of ATI envisioned will be of 72 weeks [24 weeks in AELIX-002 study + 48 weeks in current study]), followed by 24 weeks of safety follow-up after cART is resumed.

The primary objective of this study is to assess the safety and durability of viral control after AELIX-002 clinical trial intervention beyond 6 months of ATI. Furthermore, the study will collect biological samples to be stored for further investigational studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the AELIX-002 clinical trial at week 24 of ATI:

  1. Willing to continue the ATI up to 1 year.
  2. With pVL <2,000 copies/ml at week 24 of ATI on the AELIX-002 study.
  3. CD4 count ≥350 cells/mm3 at week 24 of ATI on the AELIX-002study.
  4. Willing to comply with the measures to prevent HIV transmission and reinfection required by the protocol.
  5. Available for follow-up for the planned duration of the ATI period of this study.
  6. Willing to accept blood draws and collect stool at time points specified in the Schedule of Procedures.
  7. If heterosexually active female; using an effective method of contraception (hormonal contraception, intra-uterine device

     (IUD), or anatomical sterility in self or partner1) during the ATI and until her pVL is <50 copies/ml after cART resumption.
  8. If heterosexually active male; using an effective method of contraception (anatomical sterility in self) or agree on the use of an effective method of contraception by his partner (hormonal contraception, intra-uterine device (IUD), or anatomical

     sterility1) during the ATI and until his pVL is <50 copies/ml after cART resumption.
  9. Not willing to donate blood during the study.
  10. Participants who understand the information provided, in the opinion of the investigator.

      Exclusion Criteria:

  1- Pregnancy or breastfeeding.

  2. History or clinical manifestations of any physical or psychiatric disorder which could impair the subject's ability to complete the study.

  3. Any other current or prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study.

  4. Active hepatitis B or C at week 24 of ATI on the AELIX-002 study.

  5. Risk of HIV transmission (i.e. repeated STI during the AELIX-002 ATI period or reported unprotected anal sex).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with viral remission | week 72
  Percentage of participants with viral remission, defined as plasma viral load (pVL) <50 copies/ml at 72 weeks after start of ATI.
Percentage of participants with viral control | week 72
  Percentage of participants with viral control, defined as a pVL <2,000 copies/ml at 72?weeks after start of ATI.
Time to viral detection | up to 72weeks after start of ATI
  Time to viral detection up to 72 weeks after start of ATI, defined as the time from ATI start to first occurrence of detectable pVL (≥50 copies/ml).
Time to viral rebound | up to 72 weeks after start of ATI
  Time to viral rebound up to 72 weeks after start of ATI, defined as the time from ATI start to first occurrence of ≥ 2,000 copies/ml.
Percentage of participants who remain off cART | Week 72
  Percentage of participants who remain off cART at 72 weeks after ATI start.
Time off cART | From ATI start to week 72
  Time off cART, defined as time to cART resumption from ATI start.

SECONDARY OUTCOMES:
Phenotypes characterization | From ATI start to week 72
  Different phenotypes will be characterized by the description of pVL and CD4 dynamics of each participant, and grouping according to their profile (non-rebounders, late-rebounders, post-rebound controllers, …).
Change in a score for ATI psychological impact | At weeks 24, 48 and at week 4 post cART resumption (or at the End of ATI visit in case of early withdrawal).
  Acceptability and the psychological impact of a longer ATI will be assessed by the change in a score of a questionnaire administered at weeks 24, 48 and at week 4 post cART resumption (or at the End of ATI visit in case of early withdrawal).
The proportion of participants who develop symptoms compatible with acute retroviral syndrome. | From ATI start to week 72
  The proportion of participants who develop symptoms compatible with acute retroviral syndrome.
The proportion of participants who suppress pVL to <50 copies/ml | 24 weeks after cART resumption
  The proportion of participants who suppress pVL to <50 copies/ml 24 weeks after cART resumption
The proportion of participants who develop new mutations not present in the pre-cART genotype | 24 weeks after cART resumption
  The proportion of participants who develop new mutations not present in the pre-cART genotype conferring clinically-significant resistance to antiretroviral drugs (out of the individuals not reaching viral re-suppression 24 weeks after cART resumption).
Description of participants who develop AEs related to the prime- boost regimen during this extension of ATI period. | From ATI_extension start to week 72
  Description of participants who develop AEs related to the prime-boost regimen during this extension of ATI period.

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain